CLINICAL TRIAL: NCT00713947
Title: Comparative Effectiveness of the Eradication of Helicobacter Pylori and an Inhibitor of Pump With Proton Versus Control on the Gastric Lesions Induced by the Aspirin With the Low Dose Among Patients Treated With the Long Course
Brief Title: Effectiveness of the Eradication of Helicobacter Pylori and an Inhibitor of Pump With Proton Versus Control
Acronym: Aspylori
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P051021; AOM 05114
Record Dates: First submitted 2008-06-18; First posted 2008-07-14 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Positive Helicobacter Pylori Serology; Coronary Thrombosis; Supra-aortic Artery Thrombosis
Keywords: Gastric lesions induced by low dose of aspirin; Helicobacter pylori
MeSH Terms: conditions — Coronary Thrombosis | interventions — Amoxicillin; Metronidazole; Pantoprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Amoxicillin, Clarythromycin or metronidazole,Pantoprazole,Placebo
  Interventions: Drug: during one week for the active treatments
- B (Experimental): Pantoprazole
  Interventions: Drug: Pantoprazole
- C (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Formula 515

INTERVENTIONS:
Drug: during one week for the active treatments — during one week for the active treatments placebo during 25 weeks
  Other Names: Amoxicillin; Clarythromycin or metronidazole; Pantoprazole; Placebo
  Arms: A
Drug: Pantoprazole — 6 months at 20 mg
  Arms: B
Drug: Placebo Formula 515 — 26 weeks, one tablet per day
  Arms: C

SUMMARY:
Low dose of aspirin is the main cause of gastro-duodenal ulcer. The best prevention is not definite particularly in patients without history of ulcer and infected by H. pylori.The aim of the study is to evaluate the gastric damage induced by aspirin in patients with H. pylori infection but who have any history of ulcer.

DETAILED DESCRIPTION:
The aim of the study is to compare the protective effect of H. pylori eradication versus Pantoprazole versus placebo on the gastric damage induced by low dose of aspirin. Treatment are attributed by randomisation. Patients are followed for 6 months and gastric damage are evaluated by endoscopy at the end of this period.

ELIGIBILITY:
Inclusion Criteria:

* Patients of more than 18 years old
* Coronarography or coronary imaging or supra-aortic arterial trunks ultrasound examination performed since less 7 months and having at least an arterial vascular stenosis
* Indication for aspirin treatment for at least 12 months (at the moment of the visit of inclusion) at a posology from 80 to 125 mg per day. The treatment must be prescribed since less than 7 months.
* Patient who had since less 7 month a positive Helicobacter Pylori serology.
* For the women in age to procreate, effective mode of contraception (oral contraception, surgical sterilization, coil)
* Patient having given an informed consent according to recommendation of the CPP (institutional ethical committee).

Exclusion Criteria:

* treatment by anti-coagulant, whatever its nature and its posology, by proton pump inhibitor, H2 receptor antagonists or antiacid having to be continued beyond the day of inclusion
* Treatment by methotrexate in progress or stopped since less 3 months.
* Time of more 7 months enters the beginning of the treatment by aspirin and the visit of inclusion
* Treatment by NSAID (even occasional or self medication) under or stopped since less 3 months.
* Treatment by anti-platelet drug (clopidogrel, ticlopidine, flurbiprofen, dipyridamole or antagonist of receptor GPIIb/IIIa) in progress or stopped since less than 10 days.
* Patient with a serious pathology compromising survival in the 6 month to come.
* Patient with renal or respiratory insufficiency or a hepatic pathology having a clinical repercussion.
* History of surgery of esophagus, stomach or duodenum.
* History of digestive tract bleeding or gastro-duodenal ulcer or esophagal ulcerating proven by endoscopy.
* Allergy known to clarithromycin.
* Psychiatric disorder not controlled by treatment.
* Patients all ready include in a therapeutic protocol or to be followed for 6 month.
* Alcohol consumption higher than 100gr. per day.
* Patient non suitable for participating in the protocol or to be followed for 6 month.
* History of intolerance to salicylate.
* Constitutional or acquired hemorrhagic disease
* Pregnant woman or nursing.
* Patient in emergency, people hospitalized without their assent, people without freedom, people without social health insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Measure: severity of the ulcerated gastric lesions induced by the aspirin | 6 months

SECONDARY OUTCOMES:
To measure: percentage of patients having had at least an ulcer | 6 months
To measure: the average of the ranks of lesion in antrum and corpus. | 6 months
To measure percentage of patients having had digestive clinical events | 6 months
To measure: the average of the ranks of severity of the hemorrhagic lesions and erosive lesions evaluated in antrum and corpus by two analogical scales of 150 mm | 6 months
To measure Percentage of patients having a hemorrhagic digestive of clinical expression or detected by the biological tests. | 6 months
To measure : Elements of the histopathologic score of Sydney | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Lamarque, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hotel Dieu Hospital, Paris, France